CLINICAL TRIAL: NCT05575089
Title: Pre-operative Inspiratory Muscle Training Effectiveness and Pulmonary Function in Patients Submitted to Bariatric Surgery
Brief Title: Inspiratory Muscle Training and Pulmonary Function in Patients Submitted to Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciana Chiavegato, Physiotherapist, PhD, Professor of Master's and Doctoral Programs in Physical Therapy of Universidade Cidade de São Paulo, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UNICID2021
Record Dates: First submitted 2022-09-23; First posted 2022-10-12 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2022-05

CONDITIONS: Bariatric Surgery Candidate; Muscle Weakness; Complication,Postoperative; Respiratory Muscle
Keywords: bariatric surgery; respiratory muscle strength; pulmonary function; preoperative; postoperative complications
MeSH Terms: conditions — Muscle Weakness; Postoperative Complications | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Incentive Spirometer - The Control Group (Active Comparator): The control group will receive an aerobic exercise in the cycle ergometer that will be conducted on a cycle ergometer divided into three steps: heat 5 minutes; 20 minutes with a confortable speed ( individuallyprescribed) and 5 minutes recovery. They will also perform active respiratory exercises, and incentive spirometer during 10 face-to-face physical therapy sessions. They will be instructed to do exercises with incentive spirometer at home, 3 times a day with 30 to 40 repetitions, during all preoperative period. The patients will receive a diary to note the exercises frequency.
  Interventions: Other: Aerobic exercise in cycle ergometer; Other: Deep breathing exercises
- Inspiratory muscle training - Powerbreath - The intervention group (Experimental): This intervention group will receive the same control group protocol: aerobic exercise in cycle ergometer, divided into three steps: heat 5 minutes; 20 minutes with a confortable speed ( individually prescribed) and 5 minutes recovery and active respiratory exercises ( deep inspirations associated to raise upper limbs ( 3 times of 10 repetitions each), and, in addition, inspiratory muscle training with Powerbreath during 10 face-to-face physical therapy sessions. They will be instructed to do exercises with Powerbreath at home, 3 times a day with 30 to 40 repetitions, inspiratory load: 60% of MIP ( first evaluation - protocol admission) during all preoperative period. The patients will receive a diary to note the exercises frequency.
  Interventions: Device: Inspiratory muscle training - Powerbreath; Other: Aerobic exercise in cycle ergometer; Other: Deep breathing exercises

INTERVENTIONS:
Device: Inspiratory muscle training - Powerbreath — The device "Powerbreath" is an inspiratory muscle training used to train respiratory muscles. Currently, it is one of the most used devices for the TMI, a linear load model with continuous application of inspiratory pressure throughout inspiration, in which the inspiratory regulating valve remains open while allowing an unrestricted expiration that generates resistance through a spring or of an electronic valve system, ability to offer greater load during training.
  Arms: Inspiratory muscle training - Powerbreath - The intervention group
Other: Aerobic exercise in cycle ergometer — 10 face-to-face non consecutive sessions with 30 minutes in a cycle ergometer(divided into three steps: heat 5 minutes; 20 minutes with a comfortable and supportable speed or load ( individually prescribed) and 5 minutes recovery
Other: Deep breathing exercises — Diaphragmatic exercises ( deep inspirations) associated to raise upper limbs ( 3 times - 10 repetitions each)

SUMMARY:
Obesity is defined as a body mass index greater than or equal to 30 kg / m2 and represents a public health problem that affects the world population. It is associated with a higher frequency of cardiovascular, metabolic diseases, and respiratory morbidities, which affect the quality of life of patients. Its treatment comprises different strategies, however, due the conventional treatments, surgical treatment has been the most sought after today. Objectives: To evaluate the effectiveness of preoperative inspiratory muscle training in the evolution of respiratory muscle strength in patients undergoing bariatric surgery. Methodology: Randomized clinical trial. All patients will be assessed in the pre operative period and randomized into 2 groups: control group and intervention group. The main variables are maximum inspiratory and expiratory muscle strength (MIP and MEP), peak cough flow (PCF) and pain. Control group will perform proposed respiratory physiotherapy, aerobic exercises and use of incentive inspirometry, the intervention group will perform proposed physiotherapy, aerobic exercises and use of Powerbreathe for inspiratory muscle training. Both groups will perform 10 non consecutive face-to-face physiotherapy sessions ( up 30 days before surgery). After the surgical intervention, they will be evaluated on the first and 30th postoperative days in relation to the same variables and pulmonary complications. Statistical Analysis: Sample calculation performed through a previous study: 42 patients per group. After the intervention, they will be evaluated on the second postoperative day for days of hospitalization and pulmonary complications. Statistical Analysis: Sample calculation performed through a previous study: 42 patients per group. After the intervention, they will be evaluated on the second postoperative day for days of hospitalization and pulmonary complications. Statistical Analysis: Sample calculation performed through a previous study: 42 patients per group. Categorical variables will be summarized in absolute and relative frequencies (percentages). Information regarding numerical variables will be expressed as means, standard deviations or medians, and interquartile range, depending on the distribution of the variable. All variables will be tested in relation to their distribution. To analyze the results between groups will be used the mixed linear models and for intragroup analysis, two-way ANOVA (time and group) for the following variables: MIP and MEP, PCF and pain. Expected results: Preoperative inspiratory muscle training can maintain/improve respiratory muscle strength until the moment prior to surgery, thus better preparing the patient for the condition of surgical stress, in addition to decreasing the incidence of pulmonary complications during the hospitalization period and / or in the 30 postoperative days.

DETAILED DESCRIPTION:
This is a controlled and randomized clinical trial that included 106 patients. The protocol was approved by the ethics committee (4.395.114; CAAE: 39118720.4.0000.0064).

Inclusion and exclusion criteria The sample consisted of patients for bariatric surgery from an outpatient clinic who were referred to physiotherapy by the medical team to be submitted to the preoperative protocol. The inclusion criteria are as follows: age over 18 years, body body mass index (BMI) ≥35 kg/m2, indication for elective bariatric surgery by videolaparoscopy. The patients would be excluded if they presented hemodynamic instability (systolic blood pressure [SBP] ˂ 90mmhg or reduction greater than 40mmhg; mean blood pressure [MAP] ˂ 65mmhg; tachycardia: heart rate ˃ 100bpm; altered level of consciousness; tachypnea: respiratory rate [RR] > 18rpm; and urine output: diuresis < 0.5ml/kg/hr)17. Furthermore, patients who were not release from their health insurance to undergo the surgery, were not included in the study.

Randomization Patients will be randomized into two blocks with 42 patients each, therefore two treatment groups: control and intervention groups. Randomization will be performed by a researcher not involved in the recruitment or treatment of the patients through a random draw in Excel software. Opaque sealed envelopes were used to ensure blind randomization. The envelopes will be kept in a safe place and delivered to the responsible physiotherapist after the initial assessments. Before starting the intervention, the envelope will be opened by the researcher, revealing the group strategy (control or intervention).

Assessments Preoperative procedures The patients will be evaluated clinically and demographically by the same evaluator and had their data recorded: level of physical activity (time per week); musculoskeletal pain based on the visual analogue scale (VAS)18; cough peak flow (CPF) by a peak flow meter19; dyspnea (modified Borg scale)20; maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) by a manovacuometer21; respiratory symptoms, such as dyspnea and cough; and vital signs, including systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), respiratory rate (RR), and pulse oxygen saturation (SpO2). All the patients will be submitted to a preoperative spirometry in order to exclude previous pulmonary diseases, and, at the end of the evaluation, the patients were randomized into the control group (CG) or the intervention group (IG). All patients will be underwent to 10 preoperative physiotherapy sessions, and the preoperative evaluations took place during the first and at the end of the 10th session.

Preoperative protocol The preoperative exercise protocol will be performed in both groups under a physiotherapist's supervision in 10 non-consecutive sessions in an outpatient setting twice a week, on average 30 days before the surgical procedure. The protocol consist of diaphragmatic breathing and lung re-expansion exercises, including fractional inspiration, maximum sustained inspiration and pursed lips strategy. All respiratory exercises will be performed associated with upper limb exercises and involved three sets of 10 repetitions each. Aerobic exercise will be performed on a treadmill or cycle ergometer for 20 minutes, with the load and speed set according to the individualized prescription for each patient. During the interval between the 10 sessions, the patients in both groups will be also instructed to perform standardized exercises daily at home until the moment before surgery. Pre- and postoperative instructions will be provided by the same physiotherapist that will be the responsible for the entire perioperative period. In addition to guidelines related to the surgical procedure, the patients will be instructed to perform respiratory physiotherapy according to preoperative guidance (control or intervention group) and to wear elastic socks before, during, and after surgery. All patients will be asked to keep a diary about the proposed activities.

Control group The patients will be performed all exercises in the preoperative protocol (breathing and aerobic exercises) in addition to incentive spirometry (Respiron®) in sets of 30 repetitions (level 1), 40 repetitions (level 2), or 50 repetitions (level 3) according to their weekly evolution. It will be recommended that the patients perform incentive spirometry at home, with a frequency of three times a day and an intensity as described above.

Intervention group The IMT will be associated to the same exercises offered in the preoperative protocol (breathing and aerobic exercises). It will be performed with Powerbreathe®, (Medic Plus mechanical model), with 60% of the obtained maximum inspiratory pressure in the first preoperative physical therapy evaluation. Powerbreathe®, a muscle training device, will be available to the patients, and they were instructed to also perform 30 repetitions at home three times a day.

In the immediate postoperative period, all patients will be kept for 24 hours in the intensive care unit (ICU). In addition to the guidance received about coughing, walking, and exercise practices for the lower limbs to prevent deep venous thrombosis, all patients will be performed exercises with an incentive spirometer, every hour, 30 times, and will be remained seated between intervals. As soon as possible, they will walk around the inpatient unit accompanied by the physiotherapist. Before hospital discharge (1st PO) and on the 30th postoperative day (30th PO), the patients will return to outpatient clinic to be evaluated for pain, dyspnea, MIP, MEP, CPF, and vital signs (SBP, DBP, HR, RR, and SpO2). Pulmonary complications in the period will be checked.

Statistical analysis The sample calculation was obtained from a previous study by Lloréns et al. (2015), who evaluated inspiratory muscle strength in clinically severe patients with obesity undergoing bariatric surgery after an IMT program22. A mean MIP difference of 12 (±2) cmH2O was detected between groups (sample power = 80%, alpha error = 5%, sample loss = 15%, 42 patients per group). The variables will be previously tested in relation to their distribution. Mixed linear models will be used to analyze the differences obtained between groups and to assess the intragroup evolution, a two-factor analysis of variance (ANOVA) (time and group) will be used for the following variables: MIP and MEP, CPF, and pain. Statistical Package for the Social Sciences for Windows (SPSS) version 23.0 will be used for the analysis, and a value of 5% was considered for rejection of the null hypothesis in all tests.

ELIGIBILITY:
Inclusion Criteria:

* Accept to participate in the study
* Age over 18 years
* Any gender
* Elective bariatric surgery

Exclusion Criteria:

* Mechanical ventilation for more than 48 hours after the surgical procedure

  * Hemodynamic instability at the time of the first evaluation and persistent in the evaluation after 1 hour

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Change over time in Inspiratory muscle strength - maximum inspiratory pressure (MIP) | All patients will be assessed at baseline ( protocol admission), in the 10th session of preoperative protocol ( average 30 days), 1st postoperative day ( average 7 days after the last pre op.session) and 30th postoperative day ( 30 days after surgery)
  To measure MIP, patients will be instructed to perform a maximal inspiratory effort from residual volume (RV), using a previously calibrated analog manovacuometer (range +/- 300cmH20). The highest value obtained after three repetitions will be recorded. The obtained values will be compared to the predicted values ( Predicted equations by Neder et al.)
Change over time in Expiratory muscle strength - maximum expiratory pressure (MEP) | All patients will be assessed at baseline ( protocol admission), in the 10th session of preoperative protocol ( average 30 days), 1st postoperative day ( average 7 days after the last pre op.session) and 30th postoperative day ( 30 days after surgery)
  To measure MEP, patients will be instructed to perform a maximal expiratory effort from total lung capacity (TLC) using a previously calibrated analog manovacuometer (range +/- 300cmH20). The highest value obtained after three repetitions will be recorded. The obtained values will be compared to the predicted values ( Predicted equations by Neder et al.)
Change over time in Peak Cough Flow (PCF) | All patients will be assessed at baseline ( protocol admission), in the 10th session of preoperative protocol ( average 30 days), 1st postoperative day ( average 7 days after the last pre op.session) and 30th postoperative day ( 30 days after surgery)
  For PCF measurements, you will be asked to the patients to cough with maximum effort after a deep inspiration using a peak flow meter. The highest value obtained from three repetitions will be recorded. The obtained values will be compared to the predicted values for healthy Brazilian population.

SECONDARY OUTCOMES:
Change over time in Pain | All patients will be assessed at baseline ( protocol admission), in the 10th session of preoperative protocol ( average 30 days), 1st postoperative day ( average 7 days after the last pre op.session) and 30th postoperative day ( 30 days after surgery)
  The pain will be measured by visual numeric scale (VNS). The scale ranges from 0 to 10, with 10 being the worst possible pain.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Chiavegato, PHD, Study Chair — Federal University of São Paulo
Locations (1):
- Centro de Reabilitação Stimullus, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No